CLINICAL TRIAL: NCT05055440
Title: Evaluation of Peripheral Muscle With Ultrassonografic of Critical Patients With Covid-19
Status: Completed | Type: Observational
Sponsor: University of Pernambuco (Other)
Collaborators: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Shirley Lima Campos, Associate Professor, University of Pernambuco
Other Study IDs: UFPE
Record Dates: First submitted 2021-09-20; First posted 2021-09-24 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Respiratory Infection
Keywords: SARS-CoV-2; Intensive care unit; Coronavirus; Peripheral muscle; Atrophy muscular; Uultrasound evaluation; Critically ill
MeSH Terms: conditions — Coronavirus Infections; Muscular Atrophy; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically ventilated patients with COVID-19 in the ICU: Mechanically ventilated patients with COVID-19 admitted to the intensive care unit using sedation and neuromuscular blocker

SUMMARY:
Currently, the tools available for assessing peripheral muscle dysfunction in the intensive care setting require patient collaboration. Several studies have shown that peripheral muscle ultrasound is capable of reliably detecting morphological changes in critically ill patients, in addition to contributing to the identification of patients at higher risk of prolonged complications, especially when performed daily. In this sense, a valid, non-volitional alternative capable of determining muscle mass is through ultrasound assessment. However, current studies are characterized by a lack of standardization in their protocols, which include proper positioning of limbs, transducer, clear reference points and techniques for better visualization of the assessed muscle, in addition to significant methodological defects and inadequate sample sizes. We believe that, together with a tool capable of determining muscle mass and being a safe and non-invasive method, we can contribute to a more complete assessment of these patients, exploring outcomes such as survival, length of stay in the ICU, extubation success and functional capacity. In addition to having the potential to serve as a biomarker of muscle strength during rehabilitation, given little knowledge about the long-term physical consequences of COVID-19, thus promoting a more complete assessment, exploring morphological characteristics of the peripheral muscles resulting from the hospitalization process. and assisting the physiotherapist in clinical decision making in rehabilitation.

DETAILED DESCRIPTION:
Introduction: the length of hospital stay may be associated with factors such as the need for mechanical ventilation, severity of the underlying disease, infections, use of sedation and neuromuscular blockers. In this context, the new coronavirus (SARS-CoV-2) presents itself as a group of viruses that can cause acute respiratory syndromes with mild and severe symptoms, contributing to increased hospital stays and periods of immobility. Peripheral muscle measurement through ultrasound is a topic of growing interest in the assessment of critically ill patients. Currently, this tool has been shown to be able to assess muscle dimensions and morphology during hospitalization in the intensive care unit (ICU) and can be performed at the bedside, presenting itself as a reliable inter and intraobserver method. As this tool does not depend on patient collaboration and is a non-invasive method available in most ICUs, it can provide additional information to the physical examination and clinical impression.

Objective: to evaluate the evolution of ultrasound pattern measurements in mechanically ventilated patients admitted to the ICU.

Methods: prospective cohort study that will be carried out in the ICU of the Recife Women's Hospital, located in Recife - PE, with individuals of both genders, over 18 years old, under mechanical ventilation due to suspicion or confirmation of COVID- 19. To carry out this study, the measurement of the ultrasound pattern of peripheral muscles will be performed from admission to the ICU, with follow-up on the 3rd, 5th and 7th days under mechanical ventilation. The length of stay in the ICU and mechanical ventilation, mortality in this population will also be evaluated. Clinical, laboratory, oxygenation, ventilation, respiratory system mechanics data will also be analyzed. Data will be collected and archived for analysis, which considers differences between groups with p<0.05. All ethical principles will be respected with either written Free and Consent Term by the patient or relatives at the intensive care phase or at the post ICU discharge phase.

Expected results: to contribute to a more complete assessment of these patients, exploring outcomes such as survival, length of stay in the ICU and effects of immobility on peripheral muscle mass.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both genders;
* Age group over 18 years old;
* Individuals who had a confirmed diagnosis for COVID-19 considering their positivity through the RT-PCR exam on mechanical ventilation due to acute respiratory failure

Exclusion Criteria:

- Patients with neurological impairment or known myopathies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample consisted of volunteers with COVID - 19 admitted to the SRAG ICU on mechanical ventilation due to acute respiratory failure.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Peripheral muscle thickess measured during ultrasonography | 25 minutes
  Peripheral muscle thickess expressed in centimeters
Cross-sectional area measured during ultrasonography | 10 minutes
  Cross-sectional area thickening expressed in square centimeters

SECONDARY OUTCOMES:
Murray Score (LIS) | 1 hours
  Scoring system for lung injury including hypoxemia, respiratory system compliance, chest radiographic findings and level of PEEP. The minimum value is zero and the maximum value is sixteen. The higher the score the worse outcome.
Duration of mechanical ventilation (MV days) | Through study completion, an average of 1 week
  To quantity the number of days with use of invasive mechanical ventilation in inpatients.
ICU Mortality | Through study completion, an average of 1 week
  To quantify number of living days between ICU admission and deceased status
Simplified Acute Physiological Score (SAPS3) | 10 minutes
  Scoring system applied aims to analyze the severity of the disease during the ICU stay, consisting of previous data on the health status, complications that led to hospitalization, information related to the physiological and laboratory tests during the ICU stay
Acute Physiologic and Chronic Health Evaluation II - APACHE II | 10 minutes
  Scoring system to objectively quantify disease severity and predict hospital mortality risk.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Henrique de Moura, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Physical Therapy Department, Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dall' Acqua AM, Sachetti A, Santos LJ, Lemos FA, Bianchi T, Naue WS, Dias AS, Sbruzzi G, Vieira SR; MoVe- ICU Group. Use of neuromuscular electrical stimulation to preserve the thickness of abdominal and chest muscles of critically ill patients: A randomized clinical trial. J Rehabil Med. 2017 Jan 19;49(1):40-48. doi: 10.2340/16501977-2168. PMID 28101565
- [Result] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703
- [Result] Annetta MG, Pittiruti M, Silvestri D, Grieco DL, Maccaglia A, La Torre MF, Magarelli N, Mercurio G, Caricato A, Antonelli M. Ultrasound assessment of rectus femoris and anterior tibialis muscles in young trauma patients. Ann Intensive Care. 2017 Oct 6;7(1):104. doi: 10.1186/s13613-017-0326-x. PMID 28986861
- [Result] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Result] Formenti P, Umbrello M, Coppola S, Froio S, Chiumello D. Clinical review: peripheral muscular ultrasound in the ICU. Ann Intensive Care. 2019 May 17;9(1):57. doi: 10.1186/s13613-019-0531-x. PMID 31101987
- [Result] Gruther W, Benesch T, Zorn C, Paternostro-Sluga T, Quittan M, Fialka-Moser V, Spiss C, Kainberger F, Crevenna R. Muscle wasting in intensive care patients: ultrasound observation of the M. quadriceps femoris muscle layer. J Rehabil Med. 2008 Mar;40(3):185-9. doi: 10.2340/16501977-0139. PMID 18292919
- [Result] Hammond K, Mampilly J, Laghi FA, Goyal A, Collins EG, McBurney C, Jubran A, Tobin MJ. Validity and reliability of rectus femoris ultrasound measurements: Comparison of curved-array and linear-array transducers. J Rehabil Res Dev. 2014;51(7):1155-64. doi: 10.1682/JRRD.2013.08.0187. PMID 25437305
- [Result] Joskova V, Patkova A, Havel E, Najpaverova S, Uramova D, Kovarik M, Zadak Z, Hronek M. Critical evaluation of muscle mass loss as a prognostic marker of morbidity in critically ill patients and methods for its determination. J Rehabil Med. 2018 Aug 22;50(8):696-704. doi: 10.2340/16501977-2368. PMID 30080234
- [Result] Mourtzakis M, Parry S, Connolly B, Puthucheary Z. Skeletal Muscle Ultrasound in Critical Care: A Tool in Need of Translation. Ann Am Thorac Soc. 2017 Oct;14(10):1495-1503. doi: 10.1513/AnnalsATS.201612-967PS. PMID 28820608
- [Result] Palakshappa JA, Reilly JP, Schweickert WD, Anderson BJ, Khoury V, Shashaty MG, Fitzgerald D, Forker C, Butler K, Ittner CA, Feng R, Files DC, Bonk MP, Christie JD, Meyer NJ. Quantitative peripheral muscle ultrasound in sepsis: Muscle area superior to thickness. J Crit Care. 2018 Oct;47:324-330. doi: 10.1016/j.jcrc.2018.04.003. PMID 30224027
- [Result] Parry SM, El-Ansary D, Cartwright MS, Sarwal A, Berney S, Koopman R, Annoni R, Puthucheary Z, Gordon IR, Morris PE, Denehy L. Ultrasonography in the intensive care setting can be used to detect changes in the quality and quantity of muscle and is related to muscle strength and function. J Crit Care. 2015 Oct;30(5):1151.e9-14. doi: 10.1016/j.jcrc.2015.05.024. Epub 2015 Jun 3. PMID 26211979
- [Result] Parry SM, Puthucheary ZA. The impact of extended bed rest on the musculoskeletal system in the critical care environment. Extrem Physiol Med. 2015 Oct 9;4:16. doi: 10.1186/s13728-015-0036-7. eCollection 2015. PMID 26457181
- [Result] Sarwal A, Parry SM, Berry MJ, Hsu FC, Lewis MT, Justus NW, Morris PE, Denehy L, Berney S, Dhar S, Cartwright MS. Interobserver Reliability of Quantitative Muscle Sonographic Analysis in the Critically Ill Population. J Ultrasound Med. 2015 Jul;34(7):1191-200. doi: 10.7863/ultra.34.7.1191. PMID 26112621
- [Result] Tillquist M, Kutsogiannis DJ, Wischmeyer PE, Kummerlen C, Leung R, Stollery D, Karvellas CJ, Preiser JC, Bird N, Kozar R, Heyland DK. Bedside ultrasound is a practical and reliable measurement tool for assessing quadriceps muscle layer thickness. JPEN J Parenter Enteral Nutr. 2014 Sep;38(7):886-90. doi: 10.1177/0148607113501327. Epub 2013 Aug 26. PMID 23980134
- [Result] Turton P, Hay R, Taylor J, McPhee J, Welters I. Human limb skeletal muscle wasting and architectural remodeling during five to ten days intubation and ventilation in critical care - an observational study using ultrasound. BMC Anesthesiol. 2016 Nov 29;16(1):119. doi: 10.1186/s12871-016-0269-z. PMID 27894277
- [Result] Valls-Matarin J, del Cotillo-Fuente M, Grane-Mascarell N, Quintana S. [Variation of muscle mass and weight in critical patient]. Enferm Intensiva. 2015 Jul-Sep;26(3):86-91. doi: 10.1016/j.enfi.2015.05.001. Epub 2015 Jul 9. Spanish. PMID 26165624